CLINICAL TRIAL: NCT07395141
Title: Albumin in Acute Variceal Bleeding: A Randomized Controlled Trial: ALB-AVB Trial
Brief Title: Albumin in Acute Variceal Bleeding
Acronym: ALB-AVB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King George's Medical University (Other)
Responsible Party: Principal Investigator, Sumit Rungta, Professor (Doctor), King George's Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1098/Ethics/2025
Record Dates: First submitted 2025-11-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Variceal Bleeding; Cirrhosis
Keywords: albumin; acute variceal bleed; cirrhosis; Albumin in acute variceal bleeding
MeSH Terms: conditions — Fibrosis | interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): All the participants with acute variceal bleed will be given albumin along with standard treatment
  Interventions: Drug: Albumin
- Comparator (No Intervention): This comparator group will not receive the drug.

INTERVENTIONS:
Drug: Albumin — All the participants with acute variceal bleed will be given albumin along with standard treatment
  Other Names: Albumin in acute variceal bleed
  Arms: Intervention Arm

SUMMARY:
The objective of this randomized control clinical trial is to learn the role of albumin in patients with acute variceal bleed. The trial will include all adult patients with acute variceal bleeding and cirrhosis presenting to Medical Gastroenterology department at KGMU, Lucknow, U.P. India, will include patients with age between 18-70 years and all gender.

The primary endpoint will be re-bleeding during hospitalization and at 6 weeks. Participants will be randomized in two groups, the intervention group will receive albumin for 3 days along with standard treatment and comparison group will receive on standard treatment.

DETAILED DESCRIPTION:
Albumin in acute variceal bleeding: A randomized controlled trial: ALB-AVB Trial

Introduction:

Albumin has been found to reduce mortality in patients with acute variceal bleeding in retrospective trials. However, there is no prospective data on this issue. We aim to conduct a randomized controlled trial on the role of albumin in patients with acute variceal bleeding.

Review of the literature Acute variceal bleeding is an important decompensating event in patients with cirrhosis. It is associated with 20-30% mortality in six weeks. Standard therapy with splanchnic vasoconstrictors and endoscopic band ligation is the mainstay of treatment. Previous studies have shown that albumin may decrease the mortality and re-bleeding rate in patients with AVB, however, there is no prospective data on this.

Apart from its oncotic properties albumin has different pleiotropic effects in patients with cirrhosis. It is an anti-oxidant and also binds to cytokines. Its anti-inflammatory property is responsible for reducing portal pressure and the risk of rebleeding. Currently, albumin is used in patients with acute kidney injury, spontaneous bacterial peritonitis and during large-volume paracentesis. There is also a theoretical risk of an increase in portal pressure in patients receiving albumin. The role of albumin in AVB is largely unknown. The current recommendation does not support its use in AVB however there is no strong evidence against it too. Currently, albumin has been shown to decrease mortality and decompensation in patients with cirrhosis. Large retrospective data from China have shown that albumin infusion is associated with reduced risk of rebleeding and mortality. In that study IV albumin of 40 grams/ day was associated with reduced mortality in patients with CTP-C cirrhosis. A perfectly designed RCT is warranted to explore the role of albumin in ABV.

Aim of the study:

To explore the role of albumin in patients with AVB. Study Methodology: It will be a randomised controlled trial conducted in the department of gastroenterology, KGMU Study Centre: Department of Gastroenterology, King George Medical University Lucknow Duration of the study: 6 months after the ethical approval

Sample Size Calculation:

Primary Outcome:

The primary endpoint is re-bleeding during hospitalization and at 6 weeks.

Standard Statistical Assumptions:

Expected re-bleeding rate in the control group (no albumin): 30% Expected reduction with intervention (albumin): 15% Significance level (α): 0.05 Power (1-β): 0.8

Formula for Binary Outcomes (Re-bleeding or No Re-bleeding):

n=(〖〖(Z〗_(∝/2)+Z_β)〗^2×[p_1 (1-p_1 )+p_2 (1-p_2 )])/(p_1-p_2 )^2

Where:

p1=0.30 (control event rate) p2=0.15 (intervention event rate) Zα/2=1.96 (for 95% confidence) Zβ=0.84 (for 80% power) Adding an attrition of minimum to 5% (0.05), the sample size for study obtained was that of 126 patients that is 63 patients in each arm. But for feasibility purposes it was rounded off to achieve a final sample size of 60 patients randomly allocated in each arm.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with acute variceal bleeding and cirrhosis presenting to Medical Gastroenterology department at KGMU, Lucknow, U.P. India.

Exclusion Criteria:

1. Age < 18 years and > 70 years
2. Patients with portal vein thrombosis
3. Hepatocellular carcinoma
4. Non-cirrhotic portal fibrosis
5. Extrahepatic portal vein thrombosis
6. Patients who received albumin in the last one month
7. Patients who require fresh frozen plasma
8. Patients with heart failure
9. Patients with chronic kidney disease
10. Volume overload state

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Re-bleeding rate | Six weeks (Baveno VII Consensus)
  All patients will receive vasoconstrictors after the initial hemodynamic resuscitation. Patients will receive terlipressin/ octreotide along with standard medical and endoscopic therapy.
  The intervention planned is administration of Albumin 40 mg/day and in comparison group only standard treatment will be given Re-bleeding rate in hospital and at six weeks will be measured. Time phrame is six weeks from the event.
In hospital mortality | From enrollment to death or discharge, other outcome is measured in six weeks
  All patients will receive vasoconstrictors after the initial hemodynamic resuscitation. Patients will receive terlipressin/ octreotide along with standard medical and endoscopic therapy.
  The intervention planned is administration of Albumin 40 mg per day and in comparison group only standard treatment will be given In hospital mortality in both groups will be measured Time frame is six weeks

SECONDARY OUTCOMES:
Mortality | From enrollment to 42 days (Baveno VII Consensus)
  All patients will receive vasoconstrictors after the initial hemodynamic resuscitation. Patients will receive terlipressin/ octreotide along with standard medical and endoscopic therapy.
  The intervention planned is administration of Albumin 40 mg/day and in comparison group only standard treatment will be given Mortality rate at 42 days will be measured
Need for rescue therapy | From hospitalization to need for rescue therapy within 42 days of enrollment (Baveno VII Consensus)
  All patients will receive vasoconstrictors after the initial hemodynamic resuscitation. Patients will receive terlipressin/ octreotide along with standard medical and endoscopic therapy.
  The intervention planned is administration of Albumin 40 mg/day and in comparison group only standard treatment will be given Need for rescue therapy rate will be measured during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Sumit Rungta, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Result] Wang Z, Xie YW, Lu Q, Yan HL, Liu XB, Long Y, Zhang X, Yang JL. The impact of albumin infusion on the risk of rebleeding and in-hospital mortality in cirrhotic patients admitted for acute gastrointestinal bleeding: a retrospective study of a single institute. BMC Gastroenterol. 2020 Jun 23;20(1):198. doi: 10.1186/s12876-020-01337-5. PMID 32576140
- [Result] Sarin SK, Kumar A, Angus PW, Baijal SS, Baik SK, Bayraktar Y, Chawla YK, Choudhuri G, Chung JW, de Franchis R, de Silva HJ, Garg H, Garg PK, Helmy A, Hou MC, Jafri W, Jia JD, Lau GK, Li CZ, Lui HF, Maruyama H, Pandey CM, Puri AS, Rerknimitr R, Sahni P, Saraya A, Sharma BC, Sharma P, Shiha G, Sollano JD, Wu J, Xu RY, Yachha SK, Zhang C; Asian Pacific Association for the Study of the Liver (APASL) Working Party on Portal Hypertension. Diagnosis and management of acute variceal bleeding: Asian Pacific Association for Study of the Liver recommendations. Hepatol Int. 2011 Jun;5(2):607-24. doi: 10.1007/s12072-010-9236-9. Epub 2011 Feb 19. PMID 21484145
- [Result] Guevara M, Terra C, Nazar A, Sola E, Fernandez J, Pavesi M, Arroyo V, Gines P. Albumin for bacterial infections other than spontaneous bacterial peritonitis in cirrhosis. A randomized, controlled study. J Hepatol. 2012 Oct;57(4):759-65. doi: 10.1016/j.jhep.2012.06.013. Epub 2012 Jun 23. PMID 22732511
- [Result] Cheng HC, Chang WL, Chen WY, Tsai YC, Yeh YC, Sheu BS. Intravenous albumin shortens the duration of hospitalization for patients with hypoalbuminemia and bleeding peptic ulcers: a pilot study. Dig Dis Sci. 2013 Nov;58(11):3232-41. doi: 10.1007/s10620-013-2821-8. Epub 2013 Aug 11. PMID 23934414
- [Result] Artigas A, Wernerman J, Arroyo V, Vincent JL, Levy M. Role of albumin in diseases associated with severe systemic inflammation: Pathophysiologic and clinical evidence in sepsis and in decompensated cirrhosis. J Crit Care. 2016 Jun;33:62-70. doi: 10.1016/j.jcrc.2015.12.019. Epub 2015 Dec 29. PMID 26831575
- [Result] Fernandez J, Claria J, Amoros A, Aguilar F, Castro M, Casulleras M, Acevedo J, Duran-Guell M, Nunez L, Costa M, Torres M, Horrillo R, Ruiz-Del-Arbol L, Villanueva C, Prado V, Arteaga M, Trebicka J, Angeli P, Merli M, Alessandria C, Aagaard NK, Soriano G, Durand F, Gerbes A, Gustot T, Welzel TM, Salerno F, Banares R, Vargas V, Albillos A, Silva A, Morales-Ruiz M, Carlos Garcia-Pagan J, Pavesi M, Jalan R, Bernardi M, Moreau R, Paez A, Arroyo V. Effects of Albumin Treatment on Systemic and Portal Hemodynamics and Systemic Inflammation in Patients With Decompensated Cirrhosis. Gastroenterology. 2019 Jul;157(1):149-162. doi: 10.1053/j.gastro.2019.03.021. Epub 2019 Mar 22. PMID 30905652
- See also: https://clinicaltrials.gov/study/NCT03451292 — https://clinicaltrials.gov/study/NCT03451292
- See also: https://www.medrxiv.org/content/10.1101/2024.06.12.24308846v1.full — https://www.medrxiv.org/content/10.1101/2024.06.12.24308846v1.full
- See also: https://pubmed.ncbi.nlm.nih.gov/22732511/ — https://pubmed.ncbi.nlm.nih.gov/22732511/
- See also: https://pubmed.ncbi.nlm.nih.gov/23934414/ — https://pubmed.ncbi.nlm.nih.gov/23934414/
- See also: https://pubmed.ncbi.nlm.nih.gov/21484145/ — https://pubmed.ncbi.nlm.nih.gov/21484145/
- See also: https://pubmed.ncbi.nlm.nih.gov/32576140/ — https://pubmed.ncbi.nlm.nih.gov/32576140/
- See also: https://pubmed.ncbi.nlm.nih.gov/35120736/ — https://pubmed.ncbi.nlm.nih.gov/35120736/